CLINICAL TRIAL: NCT06864455
Title: "Effects of a Relaxation Intervention on Physiological and Psychological Outcomes Among Mothers of Preterm Infants At Hospital Sultan Abdul Aziz Shah : a Within-subject Randomized Trials"
Brief Title: Breastfeeding Relaxation Intervention Among Mothers of Preterm Infants in Hospital Sultan Abdul Aziz Shah (HSAAS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: European Society of Pediatric Gastroenterology, Hepatology and Nutrition (Other)
Responsible Party: Principal Investigator, Nurul Husna Binti Mohd Shukri, Principle Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: JKEUPM-2024-205; vot 1471 (Other Grant/Funding Number: The European Society for Paediatric Gastroenterology Hepatology and Nutrition)
Record Dates: First submitted 2024-11-21; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-08

CONDITIONS: Behaviour; Psychology; Physiology; Therapy
MeSH Terms: conditions — Behavior | interventions — Culture Media

STUDY DESIGN:
Intervention Model Description: It is a "within-subject randomized trial" is a type of experimental study where each individual is exposed to more than one treatment. In this design, each participant acts as their own control, which helps to control for individual differences and reduces variability.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Guided Imagery Meditation (Experimental): Participants will need to listen to the guided imagery meditation tape that was developed by Sheri Menelli in 2004 for breastfeeding mothers as it has been successfully used before.
  Interventions: Behavioral: Guided Imagery Meditation
- Religious Recitation (Experimental): -Participants will need to listen to Surah Ar-Rahman, which will be used in this study since it has been done previously among pregnant women in the labour process.
  Interventions: Behavioral: Religious Recitation
- Infant Video with Music (Experimental): The video will be played for 10 minutes duration and mothers will need to hold the phone to look at the slide show of their infant's image and video that will be recorded by the researcher prior session
  Interventions: Behavioral: Infant Video with Music
- Distraction with News and Media (Experimental): The researcher will instruct mothers to use their phones as they did at home for 10 minutes to measure how this distraction affects the mother's physiology and psychology.
  Interventions: Behavioral: Distraction with News and Media
- Control (Experimental): No intervention but all participants will ask to sit for 10minutes . Minimum distraction will be applied.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Guided Imagery Meditation — Audio meditation by Sheri Menelli, for 10-14minutes
  Arms: Guided Imagery Meditation
Behavioral: Religious Recitation — listen to Surah Ar-Rahman for 14 minutes
  Arms: Religious Recitation
Behavioral: Infant Video with Music — 10 minutes of slides show of infant's image and video
  Arms: Infant Video with Music
Behavioral: Distraction with News and Media — 10 minutes of phone use
  Arms: Distraction with News and Media
Behavioral: Control — All participants will ask to sit for 10minutes . Minimum distraction will be applied such as minimal or no chatting.
  Arms: Control

SUMMARY:
This study is designed to compare the effects of four relaxation interventions on both physiological and psychological outcomes in lactating mothers of preterm infants. The interventions being tested include:

* Guided Imagery Meditation (GIM)
* Religious Recitation (RR)
* Infant Video with Music
* Distraction with News and Media
* A Control session

The primary objectives of the study are to evaluate and compare how these different relaxation techniques influence the physiological and psychological well-being of mothers and identify which intervention is most effective for lactating mothers who deliver prematurely.

The main research questions are:

1. How do different interventions (GIM, RR, Infant Video with Music, Distraction with Media, and Control) affect physiological and psychological outcomes when measured within the same participants?
2. Are there significant differences in physiological and psychological outcomes when participants are exposed to different interventions (GIM, RR, Infant Video with Music, Distraction with Media, and Control) within the same group?
3. Among the interventions, which one demonstrates the most beneficial effects on physiological and psychological outcomes within the same participants?

Study Design:

Each participant will be exposed to five different sessions (one for each intervention), with a gap of 1-2 days between sessions. The interventions will be administered as follows:

* Guided Imagery Meditation (GIM)
* Religious Recitation (RR)
* Infant Video with Music
* Distraction with News and Media
* A Control session

Expected Outcomes:

This study will assess the following physiological and psychological outcomes:

Physiological changes:

* Heart Rate (HR)
* Systolic Blood Pressure (SBP)
* Diastolic Blood Pressure (DBP)
* Fingertip Temperature (FT)
* Breast milk cortisol concentration

Psychological changes:

•. Perceived Relaxation

DETAILED DESCRIPTION:
The trial aims to recruit 30 mothers of premature infants who are born between 28 and 35 weeks, which falls under the categories of early and mid-preterm. Participants will be recruited among mothers aged between 18 and 49 who are non-smokers, with no medical condition that could affect breastfeeding, and also those who are not taking any psychiatric medication, and those who are not diagnosed with mental illness. This trial also aims to recruit Muslim mothers, since one of the interventions is Religious Recitation which focuses on Qur'anic verses.

The participants will be identified through recent hospital data on premature infants born between 28 to 35 weeks gestation and through a face-to-face approach. The study information sheet will be given to interested mothers. Eligible mothers will be given consent forms after assessing the inclusion and exclusion criteria for mothers and infants. The participants will be enrolled in the study and randomized using a computerized random number generator, where the participants cannot choose which intervention to test first. One person who had no contact with the participants will do randomization five times for each participant since four interventions and controls were involved.

ELIGIBILITY:
Inclusion Criteria ( Mothers)

* Malaysian women of reproductive age (18-49 years)
* Muslim
* Non-smoker
* Understand English or Malay
* Currently breastfeed their infants
* Mothers of infants born in gestational age (28 weeks- 35 weeks)
* No medical conditions that can affect infant feeding.

Exclusion Criteria:

* Taking psychiatric medication and being diagnosed with mental illness.
* Mothers are on medication that contradicts breastfeeding (eg: under medication HIV/AIDS)
* Plan to formula feed or mix feeding their infants.
* Mothers of infants with illness that could affect breastfeeding and growth (respiratory issues, gastrointestinal issues, feeding difficulties, neurological disorder, etc)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Heart Rate (BPM) | From enrollment to the end of the 5-session intervention (within 2 weeks).
  Pre- and post-measurement of heart rate in beats per minute (BPM).
Systolic Blood Pressure (SBP) | From enrollment to the end of the 5-session intervention (within 2 weeks).
  Pre- and post-measurement of systolic blood pressure in millimeters of mercury (mmHg).
Diastolic Blood Pressure (DBP) | From enrollment to the end of the 5-session intervention (within 2 weeks).
  Pre- and post- measurement of diastolic blood pressure in millimeters of mercury (mmHg).
Fingertip Temperature (FT) | From enrollment to the end of the 5-session intervention (within 2 weeks).
  Pre- and post-measurement of fingertip temperature in degrees Celsius (°C).
Breast Milk Cortisol Level | From enrollment to the end of the 5-session intervention (within 2 weeks).
  Pre- and post-measurement of cortisol levels in breast milk, typically expressed in nanograms per milliliter (ng/mL).
Perceived Relaxation (PR) | From enrollment to the end of the 5-session intervention (within 2 weeks).
  Pre- and post-measurement of perceived relaxation levels, using a 10 cm Visual Analogue Scale (VAS). The scale ranges from 0 to 10 cm, where 0 cm (on the left) represents "completely unrelaxed" and 10 cm (on the right) represents "completely relaxed." Participants will mark a point on the scale that reflects their level of relaxation at the specified time.

SECONDARY OUTCOMES:
Fat | From enrollment to the end of the 5-session intervention (within 2 weeks).
  Pre- and post- measurement of milk fat content in grams per 100 milliliters (g/100 mL)
Carbohydrate | Frame: From enrollment to the end of the 5-session intervention (within 2 weeks)
  Pre- and post- measurement of milk carbohydrate content in grams per 100 milliliters (g/100 mL).
Total energy | Frame: From enrollment to the end of the 5-session intervention (within 2 weeks)
  Pre- and post-measurement of total energy content in kilocalories per 100 milliliters (kcal/100 mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sultan Abdul Aziz Shah UPM, Serdang Selangor, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
The study results, including aggregated data, will be shared to contribute to broader scientific understanding. However, due to privacy and confidentiality concerns, individual participant data will not be shared. Only de-identified, summary-level data (e.g., group results, statistical analyses) will be made available to the public or other researchers.

REFERENCES:
- [Background] Yu J, Wells J, Wei Z, Fewtrell M. Effects of relaxation therapy on maternal psychological state, infant growth and gut microbiome: protocol for a randomised controlled trial investigating mother-infant signalling during lactation following late preterm and early term delivery. Int Breastfeed J. 2019 Dec 16;14:50. doi: 10.1186/s13006-019-0246-5. eCollection 2019. PMID 31889973
- [Background] Yu J, Wells J, Wei Z, Fewtrell M. Randomized Trial Comparing the Physiological and Psychological Effects of Different Relaxation Interventions in Chinese Women Breastfeeding Their Healthy Term Infant. Breastfeed Med. 2019 Jan/Feb;14(1):33-38. doi: 10.1089/bfm.2018.0148. Epub 2018 Oct 23. PMID 30351172
- [Background] Mohd Shukri NH, Wells JCK, Fewtrell M. The effectiveness of interventions using relaxation therapy to improve breastfeeding outcomes: A systematic review. Matern Child Nutr. 2018 Apr;14(2):e12563. doi: 10.1111/mcn.12563. Epub 2017 Nov 6. PMID 29105966
- [Background] Mohd Shukri NH, Wells J, Eaton S, Mukhtar F, Petelin A, Jenko-Praznikar Z, Fewtrell M. Randomized controlled trial investigating the effects of a breastfeeding relaxation intervention on maternal psychological state, breast milk outcomes, and infant behavior and growth. Am J Clin Nutr. 2019 Jul 1;110(1):121-130. doi: 10.1093/ajcn/nqz033. PMID 31161202
- [Background] Rafique R, Anjum A, Raheem SS. Efficacy of Surah Al-Rehman in Managing Depression in Muslim Women. J Relig Health. 2019 Apr;58(2):516-526. doi: 10.1007/s10943-017-0492-z. PMID 28900859
- [Background] Nomkin LG, Gordon I. The relationship between maternal smartphone use, physiological responses, and gaze patterns during breastfeeding and face-to-face interactions with infant. PLoS One. 2021 Oct 8;16(10):e0257956. doi: 10.1371/journal.pone.0257956. eCollection 2021. PMID 34624025
- [Background] Keith DR, Weaver BS, Vogel RL. The effect of music-based listening interventions on the volume, fat content, and caloric content of breast milk-produced by mothers of premature and critically ill infants. Adv Neonatal Care. 2012 Apr;12(2):112-9. doi: 10.1097/ANC.0b013e31824d9842. PMID 22469966
- [Background] Ak J, Lakshmanagowda PB, G C M P, Goturu J. Impact of music therapy on breast milk secretion in mothers of premature newborns. J Clin Diagn Res. 2015 Apr;9(4):CC04-6. doi: 10.7860/JCDR/2015/11642.5776. Epub 2015 Apr 1. PMID 26023551
- [Background] Dib S, Wells JCK, Fewtrell M. A within-subject comparison of different relaxation therapies in eliciting physiological and psychological changes in young women. PeerJ. 2020 May 22;8:e9217. doi: 10.7717/peerj.9217. eCollection 2020. PMID 32509467
- [Background] Holditch-Davis D, Santos H, Levy J, White-Traut R, O'Shea TM, Geraldo V, David R. Patterns of psychological distress in mothers of preterm infants. Infant Behav Dev. 2015 Nov;41:154-63. doi: 10.1016/j.infbeh.2015.10.004. Epub 2015 Oct 22. PMID 26495909